## EFFECTS OF TRIGGER POINT MASSAGE AND STRETCHING EXERCISES ON MENSTRUATION SYMPTOMS, PAIN SEVERITY, AND QUALITY OF LIFE IN PRIMARY DYSMENORRHEA

## INFORMED CONSENT FORM

This study you are participating in is an academic study, and the title is "The Effect of Trigger Point Massage and Stretching Exercises on Menstrual Symptoms, Pain Intensity, and Quality of Life in Primary Dysmenorrhea." This study aims to demonstrate that a combination of stretching exercises and trigger point therapy is more effective in treating dysmenorrhea in women. This study, conducted by the Department of Physiotherapy and Rehabilitation at the Haliç University Graduate Education Institute, will involve women between the ages of 18 and 30 who have never given birth and are diagnosed with dysmenorrhea.

If you agree to participate voluntarily in this study, Physiotherapist Zeynep İrem KAR will collect your personal information, such as your name, age, education level, and smoking status. After obtaining your full name, your surname, your education level, and your smoking history, your menstrual pain and fatigue levels, and your quality of life will be assessed using assessments such as the Visual Analog Scale (VAS), the Menstrual Symptom Scale, and the SF-36. Measurements will be made.

Before any tests are conducted, the purpose of the study will be explained, and your written consent will be obtained through an informed consent form. Trigger point massage and stretching exercises will be used in this study, and these treatments may cause muscle pain and fatigue. The expected benefits for you include a reduction in menstrual-related pain and menstrual symptoms following the use of trigger point and stretching exercises, and an improvement in attitudes toward menstruation and quality of life.

Any developments that may concern you during the study will be reported to you or your legal representative immediately. For additional information about the study or to report any problems, adverse effects, or other discomfort related to the study, you can contact Physician Zeynep İrem KAR at zeynepkar97@hotmail.com or by phone at 05312810075.

You will not be paid for your participation in this study; furthermore, no fees will be charged to you or your social security institution for any examinations, tests, or medical care services within the scope of this study. The research is not supported by any institution or organization. Participation in this research is entirely voluntary. You may refuse to participate in the research or withdraw from the research at any stage; this will not result in any penalty or hinder your benefits. The researcher may remove you from the research, with or without your knowledge, for failure to meet applicable requirements or disruptions to the study program. The results of the research will be used for scientific purposes; if you withdraw from the study or are removed by the researcher, your medical data may also be used for scientific purposes if necessary.

All your medical and identity information will be kept confidential, and your identity will not be disclosed even if the study is published. However, research audiences, investigators, ethics committees, and official authorities may access your medical information if necessary. You may also access your own medical information if you wish.

## PARTICIPANT DECLARATION

Ms. Zeynep İrem KAR informed me that this would be an academic research project and provided me with the above information regarding this research. Following this information, I was invited to participate as a "participant" in this research. If I participate in this research, I believe that the confidentiality of my information, which must remain between me and my physiotherapist, will be treated with the utmost care and respect during this research. I have been given sufficient confidence that my personal information will be meticulously protected during the use of the research results for educational and scientific purposes.

I may withdraw from the research without giving any reason during the project. (However, I am aware that it would be appropriate to notify the researchers in advance of my withdrawal to avoid causing difficulties.) I may also be excluded from the research by the researcher, provided that my medical condition is not compromised.

I assume no financial responsibility for research expenses. I will not be reimbursed.

I understand that if I encounter any problems during the research, I can reach Physician Zeynep İrem KAR at zeynepkar97@hotmail.com or 005312810075 at any time.

I am not obligated to participate in this research and may choose not to participate. I have not encountered any coercive behavior regarding my participation. If I refuse to participate, I can contact her at any time. I also know that if I refuse, it will not harm my medical care or my relationship with the physiotherapist in any way. I have fully understood all the explanations given to me. After a period of self-reflection, I have decided to complete this research project. I have decided to participate as a "participant" (subject). I accept this invitation with great pleasure and voluntarily.

A signed copy of this form will be provided to me.

## **VOLUNTEER CONSENT FORM**

I have read the text above outlining the information that must be provided to volunteers before the study. I have been given written and verbal explanations regarding these information. Under these conditions, I agree to participate in this clinical trial voluntarily and without any pressure or coercion.

Volunteer's Name-Surname:

Address: Tel.-Fax:

Date and Signature:

For those under guardianship or tutelage, the parent or guardian,

Name-Surname:

Address:

Tel.-Fax:

Date and Signature:

The researcher making the statements,

Name-Surname: Zeynep İrem KAR

Position: Physiotherapist

Tel.: 05312810075 Date and Signature: